CLINICAL TRIAL: NCT02427178
Title: MNGIE (Mitochondrial Neurogastrointestinal Encephalomyopathy) AHSCT (Allogeneic Hematopoietic Stem Cell Transplant) Safety Study
Brief Title: MNGIE Allogeneic Hematopoietic Stem Cell Transplant Safety Study
Acronym: MASS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Michio Hirano, MD (Other)
Collaborators: Cornell University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Michio Hirano, MD, Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAI1718; U54NS078059 (NIH); NCT02363881 (obsolete NCT alias)
Record Dates: First submitted 2015-02-10; First posted 2015-04-27 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Mitochondrial Neurogastrointestinal Encephalomyopathy (MNGIE)
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; MNGIE; Stem Cell transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Experimental): Hematopoietic allogeneic stem cells will be transplanted:
  HLA testing will be performed on potential stem cell donors. HLA 10/10 matched donors are eligible, however there are additional criteria that will be applied to determine an acceptable donor. Patients will receive 2 X10 6 CD34 cells/kg weight.
  Interventions: Biological: Hematopoietic Allogeneic Stem Cells

INTERVENTIONS:
Biological: Hematopoietic Allogeneic Stem Cells — HLA 10/10 matched allogeneic bone marrow cells will be infused into recipient (patient).

SUMMARY:
The purpose of this study is to find out if a stem cell transplant is safe for patients with a very rare disease. The stem cell transplant is called AHSCT (for "allogeneic hematopoetic stem cell transplantation"). The rare disease is called MNGIE (for "Mitochondrial NeuroGastroIntestinal Encephalomyopathy"). Patients with MNGIE will be transplanted with stem cells from an individual who is human leukocyte antigen (HLA) 10/10 matched. The purpose of the transplant is the production of thymidine phosphorylase.

DETAILED DESCRIPTION:
Patients who have been identified as having MNGIE by genetic testing and/or reduced thymidine phosphorylase levels will be considered for this study. The study team physician will evaluate the condition of the patient and determine if they are eligible. An HLA matched donor is necessary for transplantation. If a suitable donor is found the transplant process can proceed. The patient receives immunosuppressive therapy ( 1 week in the hospital) with subsequent IV transfer of stem cells from the donor. The patient remains in the hospital for approximately 1 month to monitor the transplant. The patient is required to attend research visits at days 0, 100, 6m, 18m and 24 m.

ELIGIBILITY:
Inclusion Criteria:

* Homozygous or compound heterozygous mutations in the TYMP gene
* Plasma thymidine level >3micromole/L
* Plasma deoxyuridine >7.5 micromole/L
* 5 to 55 years of age
* Appropriate stem cell donor (HLA 10/10 matched)
* Karnofsky performance of at least 55

Exclusion Criteria:

* Severe cognitive impairment
* Severe psychiatric illness
* Moderate to severe lung disease
* Prior episode of peritonitis due to perforated diverticula
* Prior episode of intestinal pseudo-obstruction
* Moderate to severe hepatopathy
* Moderate to severe diabetes Mellitus
* Moderate to severe cardiomyopathy
* Moderate to severe nephropathy
* Pregnancy or planning to become pregnant during study
* Hypersensitivity to E.coli derived products
* HIV disease
* Positive to anti-donor HLA DP

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
neutrophil count (cells/L) | 42 days
  engraftment success

SECONDARY OUTCOMES:
number of patient survival days | 100 days
  is the patient al
chimerism percentage | 100 days
  percent of donor cell chimerism at 100 days
micromole/l dUrd | 100 days
  level of deoxyuridine
micromole Thd | 100 days
  level of thymidine

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Yes
When applicable, we will submit a manuscript describing the results

REFERENCES:
- [Background] Halter J, Schupbach W, Casali C, Elhasid R, Fay K, Hammans S, Illa I, Kappeler L, Krahenbuhl S, Lehmann T, Mandel H, Marti R, Mattle H, Orchard K, Savage D, Sue CM, Valcarcel D, Gratwohl A, Hirano M. Allogeneic hematopoietic SCT as treatment option for patients with mitochondrial neurogastrointestinal encephalomyopathy (MNGIE): a consensus conference proposal for a standardized approach. Bone Marrow Transplant. 2011 Mar;46(3):330-337. doi: 10.1038/bmt.2010.100. Epub 2010 May 3. PMID 20436523
- [Background] Marti R, Lopez LC, Hirano M. Assessment of thymidine phosphorylase function: measurement of plasma thymidine (and deoxyuridine) and thymidine phosphorylase activity. Methods Mol Biol. 2012;837:121-33. doi: 10.1007/978-1-61779-504-6_8. PMID 22215544
- [Background] Hirano M, Nishino I, Nishigaki Y, Marti R. Thymidine phosphorylase gene mutations cause mitochondrial neurogastrointestinal encephalomyopathy (MNGIE). Intern Med. 2006;45(19):1103. doi: 10.2169/internalmedicine.45.6064. Epub 2006 Nov 1. No abstract available. PMID 17077575
- [Background] Valentino ML, Marti R, Tadesse S, Lopez LC, Manes JL, Lyzak J, Hahn A, Carelli V, Hirano M. Thymidine and deoxyuridine accumulate in tissues of patients with mitochondrial neurogastrointestinal encephalomyopathy (MNGIE). FEBS Lett. 2007 Jul 24;581(18):3410-4. doi: 10.1016/j.febslet.2007.06.042. Epub 2007 Jun 27. PMID 17612528